CLINICAL TRIAL: NCT05158803
Title: Can Lung Ultrasound Play a Competitive Role With Computed Tomography in Diagnosis and Follow up of Covid-19 Patients?
Brief Title: Lung Ultrasound in Comparison With C.T in Covid-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Amin, Sohag university, Sohag University
Other Study IDs: Soh-Med-21-12-16
Record Dates: First submitted 2021-12-12; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid 19 in acute phase
  Interventions: Radiation: ultrasound and C.T
- covid 19 follow up
  Interventions: Radiation: ultrasound and C.T

INTERVENTIONS:
Radiation: ultrasound and C.T — lung ultrasound in comparison to C.T

SUMMARY:
investigate the diagnostic ability of thoracic ultrasound in suspicious COVID-19 infection and/or COVID-19 pneumonia. Also, to compare its findings to CT and follow up these findings.

DETAILED DESCRIPTION:
ultrasound and C.T will be assessed in acute presentation of Covid 19 patients and then those patients will be reassessed again after 1 month by lung ultrasound and C.T and if ultrasound will show the same efficacy of diagnosis or not

ELIGIBILITY:
Inclusion Criteria:

* all cases of covid 19 patients

Exclusion Criteria:

* all other causes of consolidation ,ground glass fibrosis or collapse findings of C.T and ultrasound

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: covid 19 patients in acute phase and follow up after 1 and 2 months
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic ability of thoracic ultrasound for diagnosis and follow up of covid19 patients | after 1 month of acute presentation
  compare lung ultrasound with C.T finding of covid 19 patients